CLINICAL TRIAL: NCT02527967
Title: Enhanced Recovery After Surgery Protocol in Laparoscopic Surgery for Colorectal Cancer: Risk Factors for Delayed Recovery
Brief Title: ERAS in Laparoscopic Surgery for Colorectal Cancer: Risk Factors for Delayed Recovery
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Michał Pędziwiatr, Michał Pędziwiatr, MD PhD, Jagiellonian University
Other Study IDs: JagiellonianU-02
Record Dates: First submitted 2015-08-13; First posted 2015-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Colonic Neoplasms; Laparoscopy; Perioperative Care
Keywords: colorectal cancer; enhanced recovery after surgery; perioperative care; fast-track surgery; laparoscopy; minimally invasive surgery; complications
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1 (≤4 days): Group 1 consisted of patients whose hospital stay was shorter or equal to the target LOS (≤ 4 days).
- Group 1 (>4 days): In group 2 were patients whose hospital stay was longer than 4 days.

SUMMARY:
Although there is evidence for reducing complication rate and improving recovery after the implementation of Enhanced Recovery After Surgery (ERAS) protocols into colorectal surgery, most published papers include patients undergoing open resections. The aim was to analyse factors affecting recovery and length of stay (LOS) in patients after laparoscopic colorectal surgery for cancer combined with ERAS protocol.

DETAILED DESCRIPTION:
All patients were operated using laparoscopic surgery, and the perioperative care was based on pre-established ERAS protocol consisting of 13 pre and intraoperative items. Its principles and criteria for discharge from the hospital were based on the ERAS Society Guidelines.

Investigators analysed which of the factors: gender; age; BMI; ASA (American Society of Anaesthesiologists) physical status; type of surgery (colonic resection vs. rectal resection with total mesorectal excision, TME); stage of cancer; distance between the hospital and place of residence; operative time; intraoperative blood loss significantly prolong LOS (primary length of stay, excluding readmissions). Moreover, the compliance with ERAS protocol and its influence on LOS was analysed.

For the purposes of further analyses the entire group of patients was divided into 2 subgroups depending on the length of their hospital stay. On admission every patient received the information about the target length of stay of 4 days. Group 1 consisted of patients whose hospital stay was shorter or equal to the target LOS (≤ 4 days). In group 2 were patients whose hospital stay was longer than 4 days.

ELIGIBILITY:
Inclusion Criteria:

* colorectal cancer
* laparoscopic resection
* perioperative care according to ERAS principles

Exclusion Criteria:

* Patients submitted initially for open or emergency surgery
* with complex cancer who required multi-organ resection
* patients treated with endoscopic techniques using the hybrid TaTME technique (Transanal Total Mesorectal Excision)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The analysis included prospectively collected data from consecutive patients electively operated for colorectal cancer in the years 2013-2014. All patients were operated using laparoscopic surgery, and the perioperative care was based on pre-established ERAS protocol consisting of 13 items
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2013-01; Primary Completion 2014-09 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Hospital length of stay (days) | participants will be followed for the duration of hospital stay, an expected average of 4 days

SECONDARY OUTCOMES:
Compliance with ERAS protocol (%) | participants will be followed for the duration of hospital stay, an expected average of 4 days
  Compliance (%) will be calculated as the number of pre and intraoperative interventions fulfilled/13*100% (number of pre- and intraoperative protocol elements included into compliance calculations)
Complication rate (%) | up to 30 days post surgery
Readmission rate (%) | up to 30 days post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Michał Pędziwiatr, MD, PhD, Principal Investigator — 2nd Department of Surgery, Jagiellonian University, Krakow, Poland
Locations (1):
- 2nd Department of General Surgery, Krakow, Poland

REFERENCES:
- [Background] Gustafsson UO, Scott MJ, Schwenk W, Demartines N, Roulin D, Francis N, McNaught CE, Macfie J, Liberman AS, Soop M, Hill A, Kennedy RH, Lobo DN, Fearon K, Ljungqvist O; Enhanced Recovery After Surgery (ERAS) Society, for Perioperative Care; European Society for Clinical Nutrition and Metabolism (ESPEN); International Association for Surgical Metabolism and Nutrition (IASMEN). Guidelines for perioperative care in elective colonic surgery: Enhanced Recovery After Surgery (ERAS((R))) Society recommendations. World J Surg. 2013 Feb;37(2):259-84. doi: 10.1007/s00268-012-1772-0. No abstract available. PMID 23052794
- [Background] Nygren J, Thacker J, Carli F, Fearon KC, Norderval S, Lobo DN, Ljungqvist O, Soop M, Ramirez J; Enhanced Recovery After Surgery Society. Guidelines for perioperative care in elective rectal/pelvic surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. Clin Nutr. 2012 Dec;31(6):801-16. doi: 10.1016/j.clnu.2012.08.012. Epub 2012 Sep 26. PMID 23062720